CLINICAL TRIAL: NCT03915977
Title: Patterns of PTSD Over Time in Adult Intensive Care Patients - Observations From the RAPIT Trial
Brief Title: Patterns of PTSD in Adult Patients After Intensive Care
Status: Completed | Type: Observational
Sponsor: Holbaek Sygehus (Other)
Collaborators: Hillerod Hospital, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 18-000080
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2012-12

CONDITIONS: Intensive Care Unit Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Post ICU recovery program — Standardized follow up program

SUMMARY:
This study aims to describe adult patients' patterns of Post-traumatic stress disorder (PTSD) at discharge, 3, and 12 months after intensive care.

DETAILED DESCRIPTION:
The present study is a secondary analysis of the RAPIT-trial study treating data from patients on Post-traumatic stress disorder (PTDS) (Jensen et al., 2016).

Design Observational study based on data from the RAPIT trial that is a non-blinded, multicentre, parallel-group RCT conducted between December 2012-2015, at 10 intensive care units (ICUs) in four out of five regions in Denmark.

Participants Patients were consecutively recruited during the first 18 months of the study. We included Danish-speaking adults (≥18 years) who received mechanically ventilated ≥48 hours and did not meet the baseline criteria of dementia. We excluded delirious patients unable to give informed consent at randomization, or patients, who were enrolled in other studies. A total of 386 adult patients were randomized to standard care (SC) plus a nurse-led intensive care recovery program or standard care alone after ICU discharge (190 intervention, 196 SC).

Outcomes In this study, we will describe variations in patients, who experience symptoms of PTSD at ICU-discharge, 3 and 12 months after intensive care based on the data collection in the RAPIT-trial (Jensen et al., 2016). We will report trial participants' symptoms of PTSD at baseline, three months and twelve months after Intensive care using the Harvard Trauma Questionnaire (HTQ) supplemented with descriptions of patients' experiences of PTSD. Symptoms of anxiety and depression were collected at 3 and 12 months, and utilization of healthcare services including mortality were obtained from hospital charts combined with self-reported data from patients. We will use descriptive statistical methods to analyze data.

Symptoms of PTSD by HTQ-IV consisted of 17 items covering three core symptoms corresponding to DSM-IV criteria for PTSD: re-experience (5 items), avoidance (7 items), and arousal (5 items). This was supplemented by four additional items: one functional and three related to stress. We used a total score, and a cut-off of ≥40 is categorized as "positive PTSD". Symptoms of anxiety and depression were assessed using the Hospital Anxiety and Depression Scale (HADS) covering two dimensions: anxiety (7 items) and depression (7 items); subscale scores were 0-21 with higher scores reflecting greater psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Non-invasive or invasive ventilation ≥ 48 hours ( Non-ivasive ventilation (NIV) from current guidelines)
* Undiagnosed dementia

Exclusion Criteria:

* Delirium at randomization (positive CAM-ICU score)
* Participations in scientific projects which include patient interviews
* Not speaking or understanding danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients (survivors)
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2012-12-02 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Post traumatic stress disorder (PTSD) | 12 months
  Harvard Trauma Questionnaire, Range 18-72

SECONDARY OUTCOMES:
Anxiety | 12 months
  Hospital Anxiety and Depression Scale (HADS) covering anxiety (7 items) Range: 0-21
Anxiety | 3 months
  Hospital Anxiety and Depression Scale (HADS) covering anxiety (7 items) Range: 0-21
Depression | 12 months
  Hospital Anxiety and Depression Scale (HADS) covering Depression (7 items) Range: 0-21
Depression | 3 months
  Hospital Anxiety and Depression Scale (HADS) covering depression (7 items) Range: 0-21
PTSD | Baseline
  Harvard Trauma Questionnaire, Range 18-72
PTSD | 3 months
  Harvard Trauma Questionnaire, Range 18-72
PTSD | Over time at baseline, 3 and 12 months
  Change score using Harvard Trauma Questionnaire, Range 18-72
Anxiety | Over time at 3 and 12 months
  Change score Using Hospital Anxiety and Depression Scale (HADS) covering anxiety (7 items) Range: 0-21
Depression | Over time at 3 months and 12 months
  Change score using Hospital Anxiety and Depression Scale (HADS) covering depression (7 items) Range: 0-21

CONTACTS AND LOCATIONS:
Overall Officials: Janet F Jensen, Study Director — Holbaek Sygehus and Hillerod Hospital
Locations (1):
- Holbæk Hospital, Holbæk, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jensen JF, Overgaard D, Bestle MH, Christensen DF, Rattray J, Egerod I. Intervention fidelity in postintensive care follow-up consultations at ten sites in the RAPIT-trial: A mixed-methods evaluation. J Adv Nurs. 2019 Apr;75(4):862-875. doi: 10.1111/jan.13949. Epub 2019 Feb 12. PMID 30644124
- [Result] Jensen JF, Egerod I, Bestle MH, Christensen DF, Elklit A, Hansen RL, Knudsen H, Grode LB, Overgaard D. A recovery program to improve quality of life, sense of coherence and psychological health in ICU survivors: a multicenter randomized controlled trial, the RAPIT study. Intensive Care Med. 2016 Nov;42(11):1733-1743. doi: 10.1007/s00134-016-4522-1. Epub 2016 Sep 30. PMID 27695894
- See also: Homepage for project collaborators — https://posticu.wordpress.com/